CLINICAL TRIAL: NCT03378856
Title: Partnership Initiative for the Evaluation of Technological Innovation in Radiotherapy
Brief Title: Evaluation of Technological Innovation in Radiotherapy
Acronym: PERA
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 17.032
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective cohort study of patients receiving standard-care radiotherapy is paramount to a better understanding of radiation effects and longterm outcomes.

The primary objective is to determine the feasibility of establishing infrastructure to systematically collect clinical data, patient-reported outcomes, and imaging data from daily radiotherapy practice.

Secondary objectives are to provide a control cohort for comparative effectiveness research of investigational interventions through a cmRCT design; compare imaging features with clinical outcomes; understand dose-effect relationships; quantify imaging quality metrics.

DETAILED DESCRIPTION:
The study consists of an effort to develop infrastructure that will support systematic collection of data from daily radiotherapy practice. At the core, PERA is a large observational cohort study, serving as a multiple cohort randomized trial and image banking facility. It includes consent for the collection of imaging data, patient-reported outcomes, and broad randomization for studies according to the innovative cohort multiple randomized controlled trial design (cmRCT).

The basis of this design is a prospective cohort of participants receiving care as usual, who give informed consent for cohort participation.

Participants can furthermore be asked for informed consent to be randomized in future RCTs conducted within the cohort. Participants are informed that they will be offered an experimental intervention if they are randomly selected. They are also informed that they otherwise might serve as controls without being notified and that their data can be used in a trial context. For each participant in the cohort, PROs are captured at baseline and at regular intervals during follow-up. Within this cohort, multiple RCTs can be conducted. The design is especially attractive for clinical research areas with rapid evolution of technology, and for highly desired or expensive interventions.

In the first stage, at entry into the cohort, all potential participants are asked for their informed consent to participate in a cohort study and broad consent to be either randomly selected to be approached for experimental interventions or to serve as control without further notice during participation in the cohort. In a second stage, at the initiation of an RCT within the cohort, informed consent to receive the intervention is then only sought in those randomly selected for the intervention arm. At the third stage, after completion of each RCT, all cohort participants receive aggregate disclosure of trial results.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Receiving radiotherapy or brachytherapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving standard-care radiotherapy at CHUM
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Accrual rates | 2 years
  Determine feasibility of achieving high accural rates (greater than 80%) with this approach.

SECONDARY OUTCOMES:
Number of cmRCT trials activated | 2 years
  Measure if success would be the activation of 2 or more trials in the time frame.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - London Health Regional Cancer Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre de santé et de services sociaux de Laval, Laval, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHUQ, Québec, Quebec

REFERENCES:
- [Derived] Petit C, Delouya G, Taussky D, Barkati M, Lambert C, Beauchemin MC, Clavel S, Mok G, Pare AG, Nguyen TV, Duplan D, Keu KV, Saad F, Juneau D, Menard C. PSMA-PET/CT-Guided Intensification of Radiation Therapy for Prostate Cancer (PSMAgRT): Findings of Detection Rate, Effect on Cancer Management, and Early Toxicity From a Phase 2 Randomized Controlled Trial. Int J Radiat Oncol Biol Phys. 2023 Jul 15;116(4):779-787. doi: 10.1016/j.ijrobp.2022.12.055. Epub 2023 Jan 11. PMID 36639035
- [Derived] Belliveau C, Barkati M, Delouya G, Taussky D, Beauchemin MC, Lambert C, Beaulieu L, Beliveau-Nadeau D, Nicolas B, Carrier JF, Vigneault E, Menard C. Focal HDR brachytherapy boost to stereotactic radiotherapy (fBTsRT) for prostate cancer: a phase II randomized controlled trial. Radiat Oncol. 2022 Dec 9;17(1):203. doi: 10.1186/s13014-022-02173-5. PMID 36494834
- [Derived] Alley S, Jackson E, Olivie D, Van der Heide UA, Menard C, Kadoury S. Effect of magnetic resonance imaging pre-processing on the performance of model-based prostate tumor probability mapping. Phys Med Biol. 2022 Dec 13;67(24). doi: 10.1088/1361-6560/ac99b4. PMID 36223780